CLINICAL TRIAL: NCT02894515
Title: Interventional, Randomised, Open-label, Two-way Crossover, Single-dose Bioequivalence Study of Idalopirdine in Healthy Subjects Comparing the 10 mg Commercial Tablet (Test) to the 10 mg Clinical Tablet (Reference)
Brief Title: Bioequivalence Study of Idalopirdine in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn based on new efficacy data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16976A; 2016-000405-37 (EudraCT Number)
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test/Reference (Experimental): Single dose of commercial tablet Treatment A (Test) in period I. Followed by single dose of clinical tablet Treatment B (Reference) in period II. First and second dose administration will be separated by a washout period of at least 7 days
  Interventions: Drug: Idalopirdine commercial tablet (test); Drug: Idalopirdine clinical tablet (reference)
- Reference/Test (Experimental): Single dose of clinical tablet Treatment B (Reference) in period I. Followed by single dose of commercial tablet Treatment A (Test) in period II. First and second dose administration will be separated by a washout period of at least 7 days
  Interventions: Drug: Idalopirdine commercial tablet (test); Drug: Idalopirdine clinical tablet (reference)

INTERVENTIONS:
Drug: Idalopirdine commercial tablet (test) — single dose, 10 mg, oral
Drug: Idalopirdine clinical tablet (reference) — single dose, 10 mg, oral

SUMMARY:
The purpose of this study is to investigate whether 2 different tablet compositions are similar regarding absorption (uptake) in the body. One composition was used in the clinical development program and the other is intended for the market

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women with a body mass index (BMI) of >18.5 and <30 kg/m2.

Exclusion Criteria:

* pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Area under the idalopirdine plasma concentration-time curve (AUC0-t) from time zero to the last quantifiable concentration post-dose | baseline to 72 hours post-dose
Maximum observed concentration of idalopirdine (Cmax) | baseline to 72 hours post-dose

SECONDARY OUTCOMES:
Time to occurrence of Cmax (tmax) | baseline to 72 hours post-dose
Area under the idalopirdine plasma concentration-time curve (AUC0-inf) from time zero to infinity | baseline to 72 hours post-dose
Apparent elimination half-life (t1/2) | baseline to 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- GB1050, Leeds, United Kingdom